CLINICAL TRIAL: NCT02027480
Title: Antiretroviral Therapy and Inflammatory and Coagulation Biomarkers: Establishment of a Prospective Cohort, iMACS Study
Brief Title: Antiretroviral Therapy and Inflammatory and Coagulation Biomarkers: iMACS Study
Acronym: iMACS
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Wafaa Mahmoud El-Sadr, University Professor; Director, ICAP, Columbia University
Other Study IDs: AAAM2314
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: HIV (Human Immunodeficiency Virus); AIDS (Acquired Immune Deficiency Syndrome); Tuberculosis; Non-communicable Diseases (NCD)
Keywords: Antiretroviral Therapy (ART); Biomarkers; Nyanza Province; Kenya
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis; Noncommunicable Diseases

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples will be collected from study participants at 4 different points during their 12 months of participation. 15 mL of blood and 10 mL of urine will collected via venipuncture at baseline, 2 months, 6 months, and 12 months. Specimens will be retained for 10 years.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Prospective Cohort: The study will be a prospective cohort study of HIV-infected adults initiating ART at 4-8 health facilities in Nyanza Province, Kenya. Participants will be asked to take part in four visits over a 12 month period.
  At each study visit, participants will be asked questions related to demographic characteristics, medical history, including history of/recent medical conditions, family medical history, TB history and smoking status. Participants will also have their height (at baseline visit only) and weight measured for calculation of BMI and blood pressure reading. Blood and urine specimens will be collected and stored at each study visit for future testing.

SUMMARY:
The aim of this study is to develop and follow a cohort of human immunodeficiency virus (HIV)-infected adults who are starting HIV drugs at health facilities in Kenya. Blood and urine samples will be collected from all participants in order to establish a sample bank of samples in order to further the understanding of the levels of inﬂammatory biomarkers and coagulation biomarkers in African patients and the effect of taking HIV drugs on these biomarkers. This study will enroll and follow 685 men and women who are starting HIV drugs and collect blood and urine specimens from them at 4 study visits. These samples will be frozen and stored for future testing related to inﬂammatory and coagulation biomarkers.

DETAILED DESCRIPTION:
Biomarkers have been investigated as predictors of HIV disease progression, i.e. development of acquired immunodeficiency syndrome (AIDS) deﬁning diagnoses or death. There are limited data on the levels of these biomarkers among HIV-infected individuals in sub Saharan Africa and on the effect of antiretroviral therapy (ART) initiation on these levels. In addition, further work is needed to examine the association between such markers and various complications associated with HIV as well as mortality in sub Saharan Africa. The overall aim of this study is to develop a cohort of HIV-infected adults who are initiating ART at health facilities in Kenya and to establish a sample bank of plasma and urine samples in order to further the understanding of the levels of inﬂammatory biomarkers (IBM) and coagulation biomarkers (CBM) in African patients and the effect of ART initiation on these biomarkers. The study objectives are as follows:

* To recruit, establish and follow a cohort of HIV-infected individuals who are eligible for initiation of ART through 12 months
* To obtain blood and urine samples on all cohort participants at baseline, months 2, 6, and 12 for future HIV and related research
* To describe the demographic and disease characteristics of cohort participants and associations with various biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years of age
* Known to be HIV positive
* ART-naïve (with exception of prior exposure to single dose nevirapine in women)
* Documented ART eligibility based on CD4+ cell count and/or WHO staging
* Willing to provide locator information and to adhere to study procedures.
* No intention of permanently moving away from area for coming 12 months

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria outlined above
* Women who are currently pregnant
* Any condition which in the opinion of the investigators would interfere with participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort participants will be consenting HIV-infected men and women initiating ART at four to eight study sites.
Sampling Method: Non-Probability Sample
Enrollment: 685 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in mean high-sensitivity C-reactive protein (hsCRP) levels measured in mg/L | Baseline to 12 months
  Blood and urine samples of participants will be analyzed for inflammatory and coagulation biomarkers at four different times during this study to assess the change in marker levels.
Change in mean interleukin-6 (IL-6) levels measured in ng/mL | Baseline to 12 months
  Blood and urine samples of participants will be analyzed for inflammatory and coagulation biomarkers at four different times during this study to assess the change in marker levels.

SECONDARY OUTCOMES:
Prevalence (% of participants) of smoking in the study population | 12 months
  Using baseline surveys, human specimens, and other physiological measures (i.e. BP screenings), the prevalence of risk factors for non-communicable diseases will be assessed.
Prevalence (% of participants) of high BMI in the study population | 12 months
  Using baseline surveys, human specimens, and other physiological measures (i.e. BP screenings), the prevalence of risk factors for non-communicable diseases will be assessed.
Prevalence (% of participants) of cotinine in blood in the study population. | 12 months
  Using baseline surveys, human specimens, and other physiological measures (i.e. BP screenings), the prevalence of risk factors for non-communicable diseases will be assessed.
Prevalence (% of participants) of hypertension in the study population. | 12 months
  Using biomarkers, self-report, and other physiological tests (i.e. BP screenings), researchers will assess the prevalence of co-morbid conditions.
Prevalence (% of participants) of diabetes in the study population. | 12 months
  Using biomarkers, self-report, and other physiological tests (i.e. BP screenings), researchers will assess the prevalence of co-morbid conditions.
Prevalence (% of participants) of overweight/obesity in the study population. | 12 months
  Using biomarkers, self-report, and other physiological tests (i.e. BP screenings), researchers will assess the prevalence of co-morbid conditions.
Prevalence (% of participants) of tuberculosis in the study population. | 12 months
  Using biomarkers, self-report, and other physiological tests (i.e. BP screenings), researchers will assess the prevalence of co-morbid conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa M El-Sadr, MD/MPH, Principal Investigator — ICAP-NY, Columbia University
Locations (9):
- Kenya (9):
  - Ahero Sub District Hospital, Ahero, Nyanza
  - Ambira Sub District Hospital, Ambira, Nyanza
  - Awasi Mission, Awasi, Nyanza
  - Bondo District Hospital, Bondo, Nyanza
  - Nyakach District Hospital, Kisumu, Nyanza
  - Masogo Sub District Hospital, Masogo, Nyanza
  - Nyangoma Dispensary, Nyangoma, Nyanza
  - Sigomere Health Centre, Sigomere, Nyanza
  - Sondu Health Center, Sondu, Nyanza